CLINICAL TRIAL: NCT02736864
Title: Structural and Functional Repercussions of Pulmonary Tuberculosis Sequelae
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Michelle Godoy Canazza Damian, Post-graduating in Clinical Sciences of Federal University of Uberlândia; Radiologist., Federal University of Uberlandia
Other Study IDs: FUUMGCD
Record Dates: First submitted 2016-04-02; First posted 2016-04-13 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study assesses patients with cured pulmonary tuberculosis by compulsory notification data of Uberlândia (Minas Gerais state - Brazil) from 2012, 2013, 2014 and 2015. These patients will be invited by telephonic contact. After eligibility and exclusion criteria evaluation, those included will be assessed in order to know structural and functional repercussions of pulmonary tuberculosis sequelae.

DETAILED DESCRIPTION:
This study evaluates structural and functional repercussions of pulmonary tuberculosis sequelae by chest imaging (computed tomography and radiograph), functional respiratory tests (spirometry and six minute walking test) in patients with cured pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary tuberculosis with completed treatment (patients that received at least six months of treatment and with confirmed cure by negative culture and/or sputum smear, or clinical and radiological improvement after well succeed treatment);
* Treatment finalized at least one year before.

Exclusion Criteria:

* Physically impaired to perform the functional tests;
* Coexisting lung pathology (history of previous respiratory disease or clinical or radiological evidence of lung disease other than tuberculosis);
* Pregnants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cured pulmonary tuberculosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Correlation between extent of pulmonary disease by computed tomography and lung volumes by spirometry | At least one year after completion of the tuberculosis treatment
  High resolution computed tomography of the lungs will be evaluated by radiologists and the extent of pulmonary abnormalities will be score subjectively.
  Spirometry will permit assessment of lung volumes: forced expiratory volume in one second (FEV1) and forced vital capacity (FVC).

CONTACTS AND LOCATIONS:
Overall Officials: Thulio Cunha, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Clinical Hospital of Federal University of Uberlândia (Av. Pará, 1720 - Umuarama), Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No